CLINICAL TRIAL: NCT06427148
Title: Golden Breath: Feasibility and Acceptability of Biofeedback-based Virtual Reality Game for Children
Brief Title: Feasibility and Acceptability of Biofeedback-based Virtual Reality Game for Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Research assistant, Koç University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EU
Record Dates: First submitted 2024-05-15; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Population

STUDY DESIGN:
Intervention Model Description: Feedback was gathered from 10 pediatricians and nurses. Additionally, 5 inpatient children at Koç University Hospital provided their opinions on GoldenBreath, assessing ease of use, clarity, content appropriateness, sound volume, instruction clarity, game duration, and improvement suggestions. Based on feedback from 2 children suggesting more gold coins and longer game duration, options were added to adjust these elements in the game's menu.
  Stage 2: Following expert and child evaluations, a preliminary trial was conducted with 13 children at Koç University Hospital's pediatric outpatient clinic. The researcher met with children and parents ten minutes before the procedure. Children tried the game, using VR headsets and earphones during the procedure while receiving routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): To evaluate the feasibility and safety of the GoldenBreath before and after the procedure, the researchers asked the children to report their fears about the procedure. In addition, the children were asked to indicate the pain level they experienced, especially during the needle procedure. Possible missing data, withdrawal from the trial, and intervention fidelity were monitored during this process. Also, the children were monitored for fifteen minutes to see if they experienced any side effects related to the intervention.
  Interventions: Other: The biofeedback-assisted VR game "Golden Breath"

INTERVENTIONS:
Other: The biofeedback-assisted VR game "Golden Breath" — The biofeedback-assisted VR game "Golden Breath" that we presented in this study was designed to meet children's healthcare needs quickly and efficiently while reducing pain and fear during medical procedures in the pediatric population. "Golden Breath" u

SUMMARY:
The biofeedback-assisted VR game "Golden Breath" that investigators presented in this study was designed to meet children's healthcare needs quickly and efficiently while reducing pain and fear during medical procedures in the pediatric population. "Golden Breath" utilizes biofeedback techniques in a VR environment to ensure the active participation of children. By encouraging the practice of breathing techniques throughout the game, the game aims to reduce negative emotions associated with medical procedures. Through this innovative approach, investigators aim to provide new evidence supporting the effectiveness of VR and biofeedback interventions in pediatric clinical settings and ultimately improve children's overall experience during medical interventions.

DETAILED DESCRIPTION:
Children's increasing interest in phones, tablets, and computer games has led to the integration of technological interventions in pediatric healthcare services. Innovations such as telemedicine, telerehabilitation, mobile health applications, virtual reality (VR), and mobile games provide easy and accessible ways to meet children's health needs. VR, in particular, has gained popularity as a technological intervention, with numerous studies evaluating its effectiveness during children's medical procedures. Research has shown that VR use during procedures like port catheter needle insertion significantly reduces pain and fear. Similarly, VR during venipuncture has been found to positively affect children's pain, fear, and anxiety levels.

In addition to VR, integrating biofeedback technologies into VR experiences has shown positive effects on children's psychosocial outcomes. Studies on biofeedback-based VR games highlight their anxiety-reducing effects. For instance, a biofeedback-based VR game was found to reduce anxiety in children, and a neurofeedback video game, MindLight, significantly lowered anxiety levels. Another study found that a biofeedback-based video game during venipuncture helped distract children from the painful procedure, reducing their pain levels.

Combining VR and biofeedback technologies is believed to enhance intervention outcomes. Biofeedback alone may provide overly abstract or complex visual feedback, while the increased interactivity of VR boosts user engagement. Effective attention capture and active participation are crucial for developing skills and ensuring consistency through these technologies. Biofeedback in VR helps users control their physiological parameters, which is particularly beneficial for children, who can be difficult to engage effectively. These technologies can serve as effective methods for distracting children during medical procedures.

Pediatric medical procedures often cause pain, fear, and anxiety, which can persist long after the procedure and complicate treatment adherence. Therefore, controlling pain, fear, and anxiety is extremely important. Recent analyses highlight the potential of VR and biofeedback-assisted interventions to alleviate emotional distress in children. Moreover, the rise in digital engagement encourages healthcare professionals to develop new approaches to support child health in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4-12
* Applied to Koç University Hospital Pediatrics Outpatient Clinic

Exclusion Criteria:

* Children with a pain score <2 before the procedure
* Participants with previous experience with respiratory biofeedback in VR

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain-Wong-Baker Pain Assessment Scale | immediately after the intervention
  It is used to evaluate pain in children. The scale consists of six facial expressions. Facial expressions range from 0 points, "no pain-very happy" to 10 points, "unbearable pain-crying." (Wong-Baker Foundation. Home - wong-baker FACES foundation, 9.3.20. https://wongbakerfaces.org/)
Fear- Child Fear Scale | baseline and immediately after the intervention
  The scale consists of five facial expressions. In facial expressions, 0 indicates no fear, and 4 indicates severe fear (McKinley et al., 2008). The Turkish validity and reliability of the Child Fear Scale were conducted by Gerçeker and her colleagues (Özalp Gerçeker et al., 2018).
GoldenBreath Evaluation Form | During the development phase of the game
  The form created by researchers using the literature to get feedback from children about GoldenBreath consists of eight questions. It includes questions such as: Did you think the game was easy to play? Was the game suitable in terms of content? Was the sound level in the game appropriate? Was it easy for you to follow the instructions in the game? Was the use of the game sufficient in terms of time throughout the process? Is there a feature you would like to add to the game? Have you ever felt uncomfortable while playing the game?
Mobile Application Usability Scale | During the development phase of the game
  The scale was created by Hoehle (Hoehle, Aljafari, & Venkatesh, 2016), and its Turkish adaptation was made by Güler in 2019 (Güler, 2019). This tool provides information about the colors, text styles, font sizes, transitivity, application management, etc., used in the mobile application. It is used to evaluate the properties. The scale is a 7-point Likert-type measurement tool and consists of a total of 40 questions. In our study, it was used to obtain expert opinions.

IPD SHARING:
Plan to Share IPD: No